CLINICAL TRIAL: NCT02748057
Title: A Phase III, Open-label, Clinical Trial to Assess the Long Term Safety and Tolerability of MK-0653H in Japanese Patients With Hypercholesterolemia Who Have Inadequate LDL-C Control on Ezetimibe or Rosuvastatin Monotherapy
Brief Title: A Clinical Trial to Assess the Long Term Safety and Tolerability of MK-0653H in Japanese Participants With Hypercholesterolemia (MK-0653H-833)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653H-833; 163314 (Registry Identifier: JAPIC-CTI); MK-0653H-833 (Other: Merck Study Number)
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Familial Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe 10 mg + Rosuvastatin 2.5 mg (Experimental): 1 Ezetimibe 10 mg tablet and 1 Rosuvastatin 2.5 mg capsule/tablet orally, once daily for 52 weeks. If participant does not achieve low-density lipoprotein- cholesterol (LDL-C) goal after Week 12, dosage of Rosuvastatin may be increased to 5.0 mg
  Interventions: Drug: Ezetimibe; Drug: Rosuvastatin
- Ezetimibe 10 mg + Rosuvastatin 5.0 mg (Experimental): 1 Ezetimibe 10 mg tablet and 2 Rosuvastatin 2.5 mg capsules/tablets orally, once daily for 52 weeks.
  Interventions: Drug: Ezetimibe; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Ezetimibe
Drug: Rosuvastatin

SUMMARY:
The study will assess the safety and tolerability of Ezetimibe 10 mg+ Rosuvastatin 2.5 mg and Ezetimibe 10 mg+ Rosuvastatin 5.0 mg for up to 52 weeks in Japanese participants with hypercholesterolemia uncontrolled with monotherapy of Ezetimibe 10 mg or Rosuvastatin up to 5 mg.

ELIGIBILITY:
Inclusion Criteria:

* Japanese
* Outpatient with hypercholesterolemia
* Female participant who is of reproductive potential has to agree to remain abstinent or use (or partner use) two acceptable methods of birth control from date of signed informed consent to the 14 days after the last dose of study drug
* Will maintain a stable diet that is consistent with the Japan Atherosclerosis Society Guideline 2012 (JAS 2012) for prevention of atherosclerotic cardiovascular diseases for the duration of the study

Exclusion Criteria:

* Uncontrolled hypertension (treated or untreated)
* Uncontrolled type 1 or type 2 diabetes mellitus
* Homozygous Familial Hypercholesterolemia or has undergone low-density lipoprotein (LDL) apheresis
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins
* Has had a gastrointestinal tract bypass, or other significant intestinal malabsorption
* History of cancer within the past 5 years (except for successfully treated dermatological basal cell or squamous cell carcinoma or in situ cervical cancer)
* Human Immunodeficiency Virus (HIV) positive
* History of drug/alcohol abuse within the past 5 years or psychiatric illness not adequately controlled and stable on pharmacotherapy
* Consumes more than 25 g of alcohol per day
* Currently following an excessive weight reduction diet
* Currently engages in a vigorous exercise regimen (e.g.; marathon training, body building training etc.) or intends to start training during the study
* Hypersensitivity or intolerance to Ezetimibe or Rosuvastatin
* Myopathy or rhabdomyolysis with Ezetimibe or any statin
* Pregnant or lactating
* Taking any other investigational drugs and/or has taken any investigational drugs within 30 days

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teramoto T, Yokote K, Nishida C, Oshima N, Takase T. A Phase III Open-label clinical trial to assess the long-term safety of ezetimibe and rosuvastatin combination therapy in Japanese patients with hypercholesterolemia. J Clin Therapeut Med. 2018;34(11):765-82. (in Japanese) https://mol.medicalonline.jp/archive/search?jo=an9cltmd&ye=2018&vo=34&issue=11

RESULTS

PARTICIPANT FLOW:
Groups:
- Ezetimibe 10 mg + Rosuvastatin 2.5 mg: 1 Ezetimibe 10 mg tablet and 1 Rosuvastatin 2.5 mg capsule/tablet orally, once daily for 52 weeks. If participant does not achieve low-density lipoprotein-cholesterol (LDL-C) goal after Week 12, dosage of Rosuvastatin may have been increased to 5.0 mg
Period: Overall Study
Arm/Group | Ezetimibe 10 mg + Rosuvastatin 2.5 mg | Ezetimibe 10 mg + Rosuvastatin 5.0 mg
Started | 114 | 21
Completed | 109 | 19
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Participant Moved | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe 10 mg + Rosuvastatin 2.5 mg | Ezetimibe 10 mg + Rosuvastatin 5.0 mg | Total
Number analyzed (Participants) | 114 | 21 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (10.8) | 52.4 (13.3) | 57.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 9 | 70
  Male | 53 | 12 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 114 | 21 | 135
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least 1 Adverse Event (AE)
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The percentage of participants who reported at least 1 AE was summarized.
Time Frame: Up to 2 weeks post last dose of study drug (up to 54 weeks)
Population: All participants who received at least 1 dose of study drug during treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg + Rosuvastatin 2.5 mg | Ezetimibe 10 mg + Rosuvastatin 5.0 mg
Number analyzed (Participants) | 114 | 21
Percentage of Participants | 72.8 | 76.2

2. Primary Outcome: Percentage of Participants Who Had Study Drug Discontinued Due to an AE
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The percentage of participants who had study drug discontinued due to an AE was summarized.
Time Frame: up to 52 weeks
Population: All participants who received at least 1 dose of study drug during treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg + Rosuvastatin 2.5 mg | Ezetimibe 10 mg + Rosuvastatin 5.0 mg
Number analyzed (Participants) | 114 | 21
Percentage of Participants | 0.9 | 0.0

3. Secondary Outcome: Percentage Change From Baseline in Low-Density Lipoprotein-Cholesterol (LDL-C)
Description: Blood was collected at baseline (predose) and after 52 weeks of treatment to determine LDL-C levels. LDL-C was calculated using the Friedewald equation. If triglycerides (TG) exceeded 400 mg/dL (4.6 mmol/L), LDL-C was determined by beta quantification ultracentrifugation. The percentage change from baseline at Week 52 was summarized.
Time Frame: Baseline (predose) and Week 52
Population: All participants that received at least 1 dose of study drug, had baseline data for those analyses that required baseline data and had post-baseline data for endpoint.
Measure: Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Ezetimibe 10 mg + Rosuvastatin 2.5 mg | Ezetimibe 10 mg + Rosuvastatin 5.0 mg
Number analyzed (Participants) | 108 | 17
Percentage change | -33.8 [-36.9 to -30.8] | -23.9 [-29.1 to -18.6]

ADVERSE EVENTS:
Time Frame: Up to 2 weeks post last dose of study drug (up to 54 weeks)
Description: Population included all participants who received at least 1 dose of study drug during treatment period.
Arm/Group | Ezetimibe 10 mg + Rosuvastatin 2.5 mg | Ezetimibe 10 mg + Rosuvastatin 5.0 mg
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/114 | 1/21
Other Adverse Events (participants affected / at risk) | 53/114 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe 10 mg + Rosuvastatin 2.5 mg (N=114) | Ezetimibe 10 mg + Rosuvastatin 5.0 mg (N=21)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe 10 mg + Rosuvastatin 2.5 mg (N=114) | Ezetimibe 10 mg + Rosuvastatin 5.0 mg (N=21)
Gastroenteritis (Infections and infestations) | 8 (8) | 1 (2)
Nasopharyngitis (Infections and infestations) | 41 (69) | 8 (18)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Liver function test abnormal (Investigations) | 3 (3) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT02748057/Prot_SAP_000.pdf